CLINICAL TRIAL: NCT07059026
Title: Prospective Study of Thrombotic Microangiopathy (TMA) Associated With Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) In Adult Patients From Argentina
Brief Title: Thrombotic Microangiopathy (TMA) Associated With Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) In Adult Patients
Status: Recruiting | Type: Observational
Sponsor: ITAC (Instituto de Trasplantes y Alta Complejidad) (Other)
Responsible Party: Sponsor
Other Study IDs: ITAC-2024-01
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Thrombotic Microangiopathy
Keywords: Thromobotic microangiopathy; Allogeneic Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Thrombotic Microangiopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HSCT: Adults with Allogeneic Hematopoietic Stem Cell Transplantation

SUMMARY:
Thrombotic Microangiopathy (TMA) Associated with Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) is a serious complication that is associated with increased morbidity, related to multiple organ failure, with increased mortality in transplant patients. The incidence and evolution of TMA, especially in the adult population, is unclear due to the lack of early systematic screening and clear criteria for its diagnosis. For this reason, we designed this protocol to study the incidence and evolution of TMA Associated with allogeneic HSCT in adult patients from Argentina.

DETAILED DESCRIPTION:
This is a prospective multicenter non-interventional observational study that will include sites that perform routine screening using harmonized definitions and diagnostic criteria during the first 100 days post-HSCT (screening period).

All patients entering the study (HSCT accessible population), regardless of suspicion or diagnosis of TMA, will be followed every 3 months up to 12 months after transplant to evaluate secondary outcomes (follow-up period).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) undergoing allogeneic HSCT in specialized centers that, as part of their usual follow-up protocol, carry out basic screening (laboratory/clinical) for TMA and in which patients consent (within the general transplant consent), to have their data used in observational studies.
* Patients with ≥ 3/laboratory/clinical diagnostic markers of TMA in two consecutive assessments within 14 days, namely: 1-Elevated Schistocytes in peripheral blood; 2-LDH above the upper normal limit; 3-De novo thrombocytopenia or requirement for platelet transfusion; 4-De novo anemia or requirement for red blood cell transfusion; 5-High blood pressure (≥140/90); 6-Protein/creatinine ratio > 1mg/mg or proteinuria ≥ 30mg/dl in a random sample).
* Patients with suspected/diagnosed TMA who have signed the specific consent for the study.

Exclusion Criteria:

* Participation in an interventional treatment study of any therapy for TMA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) will be candidates for this study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of TMA in adult patients receiving allogeneic HSCT in specialized centers in Argentina | 100 days post-HSCT (screening period)
  The incidence of TMA will be assessed by the presence of ≥ 4/diagnostic laboratory/clinical markers present in 2 successive assessments within 14 days or if TMA is identified histologically by tissue biopsy up to day 100 post-transplant. Laboratory/clinical diagnostic markers (Harmonizing Definitions for Diagnostic Criteria and Prognostic Assessment of Transplantation-Associated published by Schoettler et al Transplant Cell Ther. 2023) are: 1-Elevated schistocytes in peripheral blood; 2-LDH above the upper limit of normal; 3-De novo thrombocytopenia or requirement for platelet transfusion; 4-De novo anemia or requirement for red blood cell transfusion; 5-High blood pressure (≥140/90); 6-Protein/creatinine ratio > 1 mg/mg or proteinuria ≥ 30 mg/dl in a random sample; 7-sC5b-9 above the upper limit of normal.

SECONDARY OUTCOMES:
Overall Survival | 3, 6, 9, 12 months (follow-up period)
  Proportion of TMA patients alive at each evaluation time frame
Non-relapse Mortality | 3, 6, 9, 12 months (follow-up period)
  Proportion of TMA patients that have died (death from any cause with exception of death due to progression or recurrence of the underlying disease) at each evaluation time frame
Proportion of patients achieving TMA response | 3, 6, 9, 12 months (follow-up period)
  TMA response is defined through the presence of response criteria (platelet count ≥ 50,000/mm3, lactate dehydrogenase < 1.5 upper limit of normal, absence of schistocytes (if present at baseline) and increase in eGFR ≥ 30% from baseline or interruption of dialysis for patients on dialysis treatment at baseline), at each evaluation time frame
Proportion of patients free of transfusion requirement | 3, 6, 9, 12 months (follow-up period)
  Assessed through the non-requirement of transfusion of red blood cells or platelets indicated for the management of TMA for ≥ 28 days, at each evaluation time frame (Transfusions required for causes other than TMA will not be considered within the evaluation of this endpoint)
Proportion of patients with high-risk TMA, | 3, 6, 9, 12 months (follow-up period)
  Assessed using the following criteria: LDH > 2 upper limit of normal; Protein/creatinine ratio > 1 mg/mg or proteinuria ≥ 30 mg/dl in a random sample; Any multi-organ dysfunction except grade 1 acute kidney injury; sC5b-9 above the upper limit of normal; Grade II-IV acute graft-versus-host disease, systemic viral or bacterial infection, evaluated at any time up to 12 months after HSCT
Proportion of patients with multiple organ dysfunction | 3, 6, 9, 12 months (follow-up period)
  Assessed through specific definitions (Schoettler et al Transplant Cell Ther. 2023)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Trasplantes de Alta Complejidad (ITAC), Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
We have not yet decided on IPD sharing

REFERENCES:
- [Background] Schoettler ML, Carreras E, Cho B, Dandoy CE, Ho VT, Jodele S, Moissev I, Sanchez-Ortega I, Srivastava A, Atsuta Y, Carpenter P, Koreth J, Kroger N, Ljungman P, Page K, Popat U, Shaw BE, Sureda A, Soiffer R, Vasu S. Harmonizing Definitions for Diagnostic Criteria and Prognostic Assessment of Transplantation-Associated Thrombotic Microangiopathy: A Report on Behalf of the European Society for Blood and Marrow Transplantation, American Society for Transplantation and Cellular Therapy, Asia-Pacific Blood and Marrow Transplantation Group, and Center for International Blood and Marrow Transplant Research. Transplant Cell Ther. 2023 Mar;29(3):151-163. doi: 10.1016/j.jtct.2022.11.015. Epub 2022 Nov 25. PMID 36442770